CLINICAL TRIAL: NCT03451058
Title: Integrated Eye Tracking and Neural Monitoring for Enhanced Assessment of Mild TBI: Clinical Optimization Study
Brief Title: Integrated Eye Tracking and Neural Monitoring for TBI: Optimization
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lynita Mullins, Department Head, Physical Medicine and Rehabilitation, United States Naval Medical Center, San Diego
Other Study IDs: NMCSD.2017.0012
Record Dates: First submitted 2017-10-03; First posted 2018-03-01 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury, eye tracking, EEG, cognition
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild TBI Group: History of head injury, Active Duty Service Member or Veteran, age 18-55, fluent in English
- Moderate to Severe TBI Group: History of head injury, Active Duty Service Member or Veteran, age 18-55, fluent in English
- Healthy Controls: No history of head injury, Active Duty Service Member or Veteran, age 18-55, fluent in English

SUMMARY:
Traumatic brain injury (TBI) is one of the most frequent injuries affecting service members. Unfortunately, current neurocognitive assessment tools are unable to reliably detect mild TBI more than a few days post- injury. Therefore, development of advanced systems for assessment and diagnosis of TBI are a top priority within Department of Defense. This project aims to evaluate a combined electroencephalography (EEG) and eye tracking system capable of assessing compromised cognitive function stemming from TBI, with the goal of enhancing operational readiness and aiding in diagnosis, improving health care and rehabilitation for affected military personnel.

DETAILED DESCRIPTION:
This study (N=100) will be a correlational study to assess cognitive function in healthy controls, individuals with mild TBI, and individuals with moderate-to-severe TBI.

In general, participants will provide demographic information, medical history, and details of their head injury. Participants will also complete a brief neuropsychological assessment to obtain an index of cognitive ability, along with the Fusion Test with eye tracking and linked EEG. MRI data may also be obtained.

ELIGIBILITY:
Inclusion Criteria:

All groups:

* Ability to use dominant hand to complete cognitive and motor tasks
* Fluent in English

Mild TBI group:

* History of mild TBI > 3 months and < 10 years prior to enrollment
* Self-report of post-concussive symptoms

Moderate-to-Severe TBI group:

- History of moderate or severe TBI > 3 months and < 10 years prior to enrollment

Exclusion Criteria:

Control group:

History of possible or confirmed brain injury

All groups:

* History of a medical condition (other than brain injury) that would be expected to affect cognitive or motor abilities (e.g. muscular dystrophy, multiple sclerosis, or psychotic disorders such as schizophrenia)
* Presence of neurological condition, such as brain tumor, brain infection, seizure, or stroke
* Presence of visual impairment that is uncorrected by glasses or contacts (including color blindness)
* Evidence of current suicidal or homicidal ideation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female service members with or without traumatic brain injury (TBI).
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
EEG | One study visit
  Spectral features and event related responses collected from scalp measurements during performance of an eye movement and working memory task.
Eye Tracking | One study visit
  Saccadic latencies measured in response to cognitive task including working memory demands.

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | One study visit
  Self-report measure of post-concussive symptoms
Trail Making Test | One study visit
  Consists of Part A and B which depends on psychomotor speed, visual search abilities, and placing demands on working memory and cognitive flexibility
Symbol Search | One study visit
  Wechsler Adult Intelligence Scale- Fourth Edition (WAIS-IV) Symbol Search measures information processing speed
Digit Span | One study visit
  WAIS-IV Digit Span including Digit Span Forward, Digit Span Backward, and Digit Span Sequencing, which measures memory span.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No